CLINICAL TRIAL: NCT01223573
Title: Newborn Pulse Oximety as a Predictor for Newborn Status and Future Outcome As Compared With the Apgar Score
Brief Title: Neonatal Pulse Oximetry Compared With Apgar Scores
Acronym: newborn O2 sat
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kern Medical Center (Other)
Responsible Party: melhem dandan, KMC
Other Study IDs: KMC1234; KMC1234 (Other: KMC)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-08

CONDITIONS: Newborns Delivered at KMC OB/GYN Department

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Apgar score is a subjective measure to assess prognosis and future outcome of a newborn. Pulse oximetry taken at 1, 5 and 10 minutes will be correlated to apgar scores in respective times in an goal to assess the usability of pulse oximetry as an added tool in determining the newborn prognosis

ELIGIBILITY:
Inclusion Criteria:

Newborns delivered vaginaly or by C-section at Kern Medical Center labor and delivery ward

Exclusion Criteria:

known cardiopulmonary disease of the newborn

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newborns delivered at KMC OBGYN dept
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Estimated)